CLINICAL TRIAL: NCT02144597
Title: The Effect of a 2-week vs. 6-week Low-calorie Diet (LCD) Followed by Roux-en-Y Gastric Bypass (RYGB) on Body Composition and Surgery Outcomes in Obese Humans: a Dietary Intervention and Magnetic Resonance Imaging Study
Brief Title: Low-calorie Diet and Body Composition Prior to Roux-en-Y Gastric Bypass
Acronym: LCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Cambridge Weight Plan Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CRO1668
Record Dates: First submitted 2014-05-09; First posted 2014-05-22 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Morbid Obesity; Liver Fat
Keywords: morbid obesity; gastric bypass; bariatrics; diet; caloric restriction; liver fat; appetite
MeSH Terms: conditions — Obesity, Morbid; Fatty Liver | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2-week LCD and Roux-en-Y gastric bypass (RYGB) (Active Comparator): A 2-week liquid formula low-calorie diet (LCD) will be administered for 2 weeks prior to Roux-en-Y gastric bypass. The diet will provide 800kcal per day in the form of powdered milkshakes and soups
  Interventions: Dietary Supplement: Liquid formula low-calorie diet (LCD); Procedure: Roux-en-Y gastric bypass (RYGB)
- 6-week LCD (Active Comparator): A 6-week liquid formula low-calorie diet (LCD) will be administered for 6 weeks prior to Roux-en-Y gastric bypass. The diet will provide 800kcal per day in the form of powdered milkshakes and soups
  Interventions: Dietary Supplement: Liquid formula low-calorie diet (LCD)
- Control diet (Other): 1000 calorie diet
  Interventions: Procedure: Roux-en-Y gastric bypass (RYGB); Other: Control diet

INTERVENTIONS:
Dietary Supplement: Liquid formula low-calorie diet (LCD) — The liquid formula low-calorie diet (LCD) will provide 800kcal/day from powdered milkshakes and soups. The diet will be provided by Cambridge Weight Plan.
  Other Names: LCD; LED; Cambridge Weight Plan
  Arms: 2-week LCD and Roux-en-Y gastric bypass (RYGB); 6-week LCD
Procedure: Roux-en-Y gastric bypass (RYGB) — Participant went through Roux-en-Y gastric bypass (RYGB) surgery
  Arms: 2-week LCD and Roux-en-Y gastric bypass (RYGB); Control diet
Other: Control diet
  Arms: Control diet

SUMMARY:
Losing weight before undergoing Roux-en-Y gastric bypass (RYGB) surgery may reduce liver fat content and size thereby improving surgical outcomes. This study aims to investigate whether a 2-week or 6-week pre-operative liquid formula low-calorie diet (LCD) reduces liver fat further than a conventional food diet prior to RYGB using magnetic resonance imaging (MRI). The hypothesis is that the 2-week and 6-week liquid formula LCD will reduce liver fat further than the conventional food pre-operative diet.

DETAILED DESCRIPTION:
The morbidly obese subjects (BMI higher then 40 kg/m2) were randomised and assessed at baseline (week 0). After 2 weeks on a low-calorie diet (LCD), participants underwent either Roux-en-Y gastric bypass (RYGB) or continued with a LCD for 4 weeks.The participants will reassess at week 6.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing Roux-en-Y gastric bypass at Imperial Weight Centre
* aged 18 to 60 years
* boby mass index of 35 to 55 kg/m2

Exclusion Criteria:

* Claustrophobia
* Pacemaker, metal implant, clips, implanted device, shrapnel or bullets, metal in eyes that precludes magnetic resonance imaging
* Current pregnancy or breast feeding for females (as determined by a pregnancy test)
* A full term pregnancy within the last year for females
* Treatment with any medication that might affect the study outcomes
* Haemorrhagic disorders and anticoagulant treatment
* History of cancer, excluding skin cancer
* History of severe or multiple allergies, severe adverse drug reaction or leucopenia
* Smokers
* Regular drinkers of more than three units of alcohol daily
* History of, or current evidence of, abuse of alcohol or any drug substance, licit or illicit
* Regular intake of over-the-counter (OTC) medication (other than the occasional paracetamol/aspirin)
* Poor compliers or subjects unlikely to commit to the 26 week study duration
* Blood donation within the 12 week period before the initial study dose
* Use of monoamine oxidase inhibitors (MAOIs) as anti depressant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Gary S Frost, RD PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical research facility, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bottin JH, Balogun B, Thomas EL, Fitzpatrick JA, Moorthy K, Leeds AR, Bell JD, Frost GS. Changes in body composition induced by pre-operative liquid low-calorie diet in morbid obese patients undergoing Roux-en-Y gastric bypass. Obesity reviews (March 2014), 15 (suppl 2): 129-176. (T5:S24.05). doi: 10.1111/obr.12151

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Diet: 1000 calorie diet
  Roux-en-Y gastric bypass (RYGB): Participant went through Roux-en-Y gastric bypass (RYGB) surgery
  Control diet
Period: Overall Study
Arm/Group | 2-week LCD and Roux-en-Y Gastric Bypass (RYGB) | 6-week LCD | Control Diet
Started | 10 | 10 | 10
Completed | 4 | 6 | 6
Not Completed | 6 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Numbers are not the same between the flow chart, the baseline results and some outcomes because depending on the variable measured, there are more or less patients. Forexemple, for some variables there might be missing data or a missing timepoint (baseline, visit 2, 3 or 4), For example, 30 were initially enrolled, 24 had data available after the baseline visit, 21 had MRI liver data at visit 3 (1 motnh post surgery) and 16 had MRI liver data at 6 months.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-week LCD and Roux-en-Y Gastric Bypass (RYGB) | 6-week LCD | Control Diet | Total
Number analyzed (Participants) | 9 | 8 | 7 | 24
Age, Continuous [Geometric Mean (Inter-Quartile Range); unit: years] | 40 [30 to 53] | 46 [36 to 60] | 40 [28 to 56] | 42 [36 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 5 | 19
  Male | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Intra-hepatocellular Lipid Content (IHCL) Following the Pre-operative Diet
Description: Intra-hepatocellular lipid content will be measured by magnetic resonance spectroscopy
Time Frame: at 2 weeks or 6 weeks depending on group
Population: The numbers are not the same because depending on the variable measured (some might have missing data) and its timepoint (baseline, visit 2, 3 or 4), there are more or less patients. For example, 29 were initially enrolled, 24 had data available after the baseline visit, 21 had MRI liver data at visit 3 (1 motnh post surgery) and 16 had MRI liver data at 6 months.
Measure: Mean (Standard Error); unit: percentage of change in IHCL
Arm/Group | 2-week LCD and Roux-en-Y Gastric Bypass (RYGB) | 6-week LCD | Control Diet
Number analyzed (Participants) | 9 | 8 | 6
percentage of change in IHCL | 40.0 (7.1) | 67.4 (9.1) | 0.1 (8.3)

2. Secondary Outcome: Change in Intra-hepatocellular Lipid Content (IHCL) Following Roux-en-Y Gastric Bypass
Description: Intra-hepatocellular lipid content (IHCL) will be compared between groups at 1 month following Roux-en-Y gastric bypass
Time Frame: at 1-month following Roux-en-Y gastric bypass
Measure: Mean (Standard Error); unit: percentage change in IHCL
Arm/Group | 2-week LCD and Roux-en-Y Gastric Bypass (RYGB) | 6-week LCD | Control Diet
Number analyzed (Participants) | 8 | 7 | 6
percentage change in IHCL | 31.8 (13.4) | 57.8 (11.9) | 26.4 (15.1)

3. Secondary Outcome: Change in Intra-hepatocellular Lipid Content (IHCL) Following Roux-en-Y Gastric Bypass
Description: Intra-hepatocellular lipid content (IHCL) will be compared between groups at 6 months following Roux-en-Y gastric bypass
Time Frame: at 6 months following Roux-en-Y gastric bypass
Measure: Mean (Standard Error); unit: percentage change in IHCL
Arm/Group | 2-week LCD and Roux-en-Y Gastric Bypass (RYGB) | 6-week LCD | Control Diet
Number analyzed (Participants) | 4 | 6 | 6
percentage change in IHCL | 69.8 (16.5) | 88.1 (3.5) | 83.0 (8.3)

4. Secondary Outcome: Complexity of Surgery
Description: Complexity of surgery will be assessed by the surgeon at the time of surgery (either after 2 weeks for the Control group and 2-week LCD group or after 6 weeks for the 6-week LCD group) The complexity of the surgery was assessed through a score on a complexity scale based on questionnaires previously published by Anders Thorell"s and David Edholm"s groups (Edholm et al., 2011, Van Nieuwenhove et al., 2011). The scores (1-5) for 7 variables: exposure, bleeding, difficulty in dissection, difficulty in reconstruction, surgical judgment, technical demand and psychological stress were combined into a complexity of surgery score with a minimum of 7 (very little complexity) and a maximum of 35 (very high complexity).
Time Frame: at the time of surgery
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | 2-week LCD and Roux-en-Y Gastric Bypass (RYGB) | 6-week LCD | Control Diet
Number analyzed (Participants) | 7 | 6 | 5
scores on a scale | 12 (5) | 13 (3) | 12 (4)

5. Secondary Outcome: Operative Time
Description: The operative time will be recorded at the time of surgery by the operating surgeon (either after 2 weeks for the Control group and 2-week LCD group or after 6 weeks for the 6-week LCD group)
Time Frame: at the time of surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 2-week LCD and Roux-en-Y Gastric Bypass (RYGB) | 6-week LCD | Control Diet
Number analyzed (Participants) | 7 | 6 | 5
minutes | 86 (13) | 72 (8) | 72 (6)

ADVERSE EVENTS:
Time Frame: From baseline until visit 4 at 6 months post surgery
Arm/Group | 2-week LCD and Roux-en-Y Gastric Bypass (RYGB) | 6-week LCD | Control Diet
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes